CLINICAL TRIAL: NCT06501586
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of SGB-3908 After a Single Administration in Healthy Subjects and Mildly Hypertensive Subjects
Brief Title: Study of SGB-3908 in Healthy Subjects and Mildly Hypertensive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-3908-001
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertension,Essential
Keywords: healthy; mildly hypertensive
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGB-3908 (Experimental)
  Interventions: Drug: SGB-3908
- SGB-3908-Matching placebo (Placebo Comparator)
  Interventions: Other: SGB-3908-Matching placebo

INTERVENTIONS:
Drug: SGB-3908 — SGB-3908 for sc injection
  Arms: SGB-3908
Other: SGB-3908-Matching placebo — Normal saline (0.9% NaCl) matching volume of SGB-3908 doses will be administered
  Arms: SGB-3908-Matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) effects of SGB-3908 in healthy subjects and mildly hypertensive subjects. The study will be a single ascending dose (SAD) phase.

ELIGIBILITY:
Inclusion Criteria:

* Has body mass index (BMI) ≥18 and ≤30 kg/m^2 and has bodyweight ≥ 50 kg;
* Has Systolic blood pressure (SBP) ≥100 mmHg and ≤150 mmHg and diastolic blood pressure (DBP) ≥65 mmHg and ≤95 mmHg at screening;

Exclusion Criteria:

* Has mental illness, liver and kidney disease, gastrointestinal disease, nervous system disease, or other related systemic diseases that affect the trial;
* Has a history of hospitalization or other clinically significant diseases within 1 month before screening, major surgery within 6 months before screening, or other unstable conditions judged by the investigator;
* Has a history of orthostatic hypotension or syncope;
* Patients with clinically significant abnormalities confirmed by physical examination, 12-lead electrocardiogram, laboratory tests, etc., or those who meet any of the following conditions during screening need to be excluded:

  1. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin higher than 1.5× upper limit of normal (ULN)
  2. Serum creatinine (Cr) higher than ULN
  3. Serum potassium higher than 5 mmol/L
  4. QT/QTc interval prolongation during screening (QTcF>450 ms)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to approximately 12 months

SECONDARY OUTCOMES:
Change from Baseline in Blood Angiotensinogen (AGT) Level | up to approximately 12 months
Maximum Observed Plasma Concentration (Cmax) of SGB-3908 and of Potential Metabolites | Up to Day 3
Area Under the Concentration-time Curve (AUC) of SGB-3908 and of Potential Metabolites | Up to Day 3
Number of Participants With Anti- SGB-3908 Antibodies | up to approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided